CLINICAL TRIAL: NCT05179343
Title: Sham Controlled RCT Evaluating the Safety, Acceptability and Efficacy of Autonomic Neuromodulation Using Trans-cutaneous Vagal Stimulation in Uncontrolled Hypertensive Patients: a Pilot Study
Brief Title: SCRATCH-HTN Study: Evaluating Autonomic Neuromodulation Using Trans-cutaneous Vagal Stimulation in Hypertensive Patients
Acronym: SCRATCH-HTN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Health Innovation Oxford and Thames Valley (Oxford AHSN) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2358563
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Uncontrolled Hypertension; High Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomised at the baseline visit to either the active (tAN) or sham (sham-tAN) device arm of the trial at a ratio 2:1 ratio.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active arm (Experimental): Participants in this arm will receive the active AffeX-CT device.
  Interventions: Device: Active AffeX-CT device
- Sham arm (Sham Comparator): Participants in this arm will receive the sham (inactive) AffeX-CT device.
  Interventions: Device: Sham AffeX-CT device

INTERVENTIONS:
Device: Active AffeX-CT device — (Trans-cutaneous Autonomic Neurostimulation) tAN treatment will be administered using AffeX-CT device (a device based on a totally TENS unit). AffeX device comprises of a battery-operated control unit, two electrode pairs arranged on ear clips and connected to the control unit with electrical leads. The AffeX device generates an electrical signal that is used to stimulate the nerves that naturally control the output from the sympathetic nervous system.
  Arms: Active arm
Device: Sham AffeX-CT device — Sham Totally TENS device. The device is identical to the active device used in the study, but its only purpose is to act as a placebo. The ear-clip electrodes have been modified so that the electric current is not transmitted to the participant.
  Arms: Sham arm

SUMMARY:
This is a pilot, sham-controlled, double blind, single-site device clinical trial designed to evaluate the safety, acceptability and efficacy of non-invasive autonomic neuromodulation in a cohort of 63 adult patients with uncontrolled high blood pressure.

DETAILED DESCRIPTION:
SCRATCH-HTN trial is a randomised sham-controlled study designed to evaluate the safety, acceptability, and efficacy of trans-cutaneous autonomic neurostimulation (tAN) in a cohort of uncontrolled medicated hypertensive patients.

SCRATCH-HTN trial is designed to test the hypothesis that tAN treatment is safe and acceptable to the patient, improves the control of blood pressure in hypertension and sense of well-being amongst those who are receiving the active treatment as compared to those on sham treatment.

The study will recruit 63 patients with systemic arterial hypertension (male and female aged ≥18 years) who are receiving between one and three oral antihypertensive medications and remain hypertensive with blood pressure (BP) above target levels detailed below in the eligibility criteria. The participants will be randomly allocated to the active (tAN) or sham (sham-tAN) arms of the trial on 2:1 basis, respectively.

The total treatment duration is 12 weeks. Self-administration of 30 min of tAN or sham stimulations once per day for the first two weeks, and then once every week for the rest of the trial period.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has given written informed consent.
2. Participant has sufficient knowledge of the English language to be able understand the participant information sheet and trial materials including outcome assessments.
3. Participant is aged ≥18 years and <80 years at the time of screening visit.
4. Participant is taking between 1 to 4 antihypertensive medications (inclusive) at time of screening and baseline (randomisation) visit and is willing to adhere to no change in medication during the trial until end of the trial visit (visit 5). (NB. Participant on only one antihypertensive medication should be taking that medication for at least six weeks prior to the screening visit).
5. Participant has confirmed diagnosis of hypertension.
6. Participant meets BP criteria:

   • 24-hour ambulatory BP monitoring (ABPM) at either screening visit or baseline (randomisation) visit, with mean daytime SBP of ≥135 mmHg and <170 mmHg and mean daytime DBP of ≥85 mm Hg and <115 mmHg (N.B. By default, Ambulatory Blood Pressure Monitoring [ABPM] at screening visit will be used at baseline visit. However, if there has been an addition of new medication after participants screening visit, 24-hour ABPM must be repeated at baseline visit).
7. Participant has one or more of the following associated conditions:

   1. Obesity: BMI >30 or waist circumference >94 cm (men) or > 80cm (women). (NB. For participants of South-East Asian/Chinese/Japanese origin these cut-offs are >90 cm (men) or >80 cm (women)).
   2. Type 2 diabetes - controlled or sub-optimally controlled (HbA1c ≤8.5% or ≤69 mmol/mol) on diet and/ or medications except insulin.
   3. Heart rate (average) ≥70 bpm at screening or baseline (randomisation) visit (measurement taken after 5 minutes of rest in a seated position and when finger probe has been placed for a minimum of 30 seconds thereafter) or a heart rate (average) ≥60 bpm at screening or baseline (randomisation) visit if the patient is taking beta-blocker medication.
   4. HbA1c ≥42 mmol/mol or fasting blood glucose (if available) ≥5.6 mmo/L AND either low HDL cholesterol (≤1.03 mmol/L for men and ≤1.29 mmol/L for women) or high triglyceride (triglycerides ≥1.7 mmol/L)
   5. Both low HDL cholesterol (≤1.03 mmol/L for men and ≤1.29 mmol/L for women) AND high triglyceride (triglycerides ≥1.7 mmol/L)
   6. Diagnosed or known case of polycystic ovarian syndrome.
8. Female participants of child-bearing potential (all those below 55 years except if they are surgically sterile, meaning they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy, or formally diagnosed by their doctors to be post-menopausal) must agree to use the acceptable methods of contraception from the time of consent until last follow up visit.
9. Participant is able to communicate satisfactorily with the Investigator and Investigation Site staff, and to participate in, and comply with all clinical study requirements.
10. Participants agrees to have all trial procedures performed and is able and willing to comply with all trial visits and protocol requirements.

Exclusion Criteria:

1. Participant is unable and unwilling to use the AffeX-CT device daily.
2. Participant has a small tragus (ie. the size or shape of the tragus is such that it doesn't allow the application of the ear-clips of the AffeX-CT device for a sustained period of time).
3. Participant has a piercing on the tragus of the ear.
4. Participant is diagnosed with atrial fibrillation or other form of cardiac arrhythmia
5. Participant is known to have chronic kidney disease (CKD) stage 3b or higher or had eGFR <45 ml/min/1.73 m2 in last three months prior to baseline (randomisation) visit.
6. Participant has type 1 diabetes mellitus.
7. Participant has type 2 diabetes mellitus on Insulin or those on oral antidiabetic medications with poor glycaemic control defined as HbA1c above 8.5% (or >69 mmol/mol).
8. Participant has a history of falls or symptoms of orthostatic hypotension in the last 3 months prior to baseline (randomisation) visit.
9. Participant is pregnant, nursing or planning to become pregnant within the next 6 months.
10. Participant suffers from chronic pain and has taken anti-inflammatory drugs for two or more days per week over the last month prior to baseline (randomisation) visit.
11. Participant has clinically significant or symptomatic hypertension-mediated target organ damage such as severe heart failure with NYHA 4, end stage renal damage, medically diagnosed/imaging proven stroke, symptomatic peripheral vascular disease, or severe retinopathy.
12. Participant has a history of stable or unstable angina or had an acute coronary event within 3 months prior to baseline (randomisation) visit or had a myocardial infarction within the last six months of enrolment prior to baseline (randomisation) visit.
13. Participant has a history of renal denervation within last 1 year prior to baseline (randomisation) visit.
14. Participant has a therapeutic implantable electronic/electrical device such as pacemaker, implantable cardioverter-defibrillators (ICDs), implanted vagal stimulators.
15. Participant has history of hospitalization (> 24 hour) for heart failure, or cerebrovascular accidents, or history of stroke diagnosed based on imaging or evidence of specialist diagnosis or any other indirect evidence such as discharge summary or clinical letter (at any time in the past).
16. Participant has mean daytime ABPM pulse pressure ≥ 80 mmHg at screening or baseline (randomisation) visit.
17. Participant has a heart rate <50 bpm at screening or baseline (randomisation) visit (measurement taken after 5 minutes of rest in a seated position and when finger probe has been placed for a minimum of 30 seconds thereafter).
18. Participant has auricular dermatitis.
19. Participant has postural hypotension, defined as a fall > 20mmHg in SBP on standing at 3 minutes (compared with sitting).
20. Participant has a history of hospitalization for hypertensive emergency or urgency in the last six months of enrolment prior to baseline (randomisation) visit.
21. Participant is identified as unsuitable to participate by the CI/Co-Investigator(s) and/or Investigation site team for another reason (e.g., for other medical reasons, laboratory abnormalities, limited life expectancy, etc.).
22. Participants with history of epilepsy and are currently on anti-epileptic medication or those who are not on any anti-epileptic medication but have history of a seizure within last 10 years.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2025-09-08 (Actual)

PRIMARY OUTCOMES:
Change in average daytime ambulatory Systolic Blood Pressure (SBP) from baseline to the end of treatment. | from baseline to 3 months
  Daytime SBP values will be obtained with 24hr ABPM

SECONDARY OUTCOMES:
Change in average daytime ambulatory SBP and Diastolic Blood Pressure (DBP) from baseline and 1 month. | from baseline to 1 month
  Daytime ambulatory SBP values will be obtained with 24hr ABPM
Change in average daytime ambulatory DBP from baseline to the end of treatment. | from baseline to 3 months
  Daytime ambulatory DBP values will be obtained with 24hr ABPM
Controlled BP at the end of treatment defined as mean daytime ambulatory SBP<135 mmHg and mean daytime ambulatory DBP<85 mmHg. | from baseline to 3 months
  Daytime ambulatory SBP and DBP will be obtained with 24hr ABPM
Change in average 24-hour ambulatory SBP and DBP from baseline to the end of treatment. | from baseline to 3 months
  Daytime ambulatory SBP and DBP will be obtained with 24hr ABPM
Change in average office SBP and DBP from baseline to 1 month, and from baseline to the end of treatment (3 months). | baseline to 1 month and baseline to 3 months
  Daytime ambulatory SBP and DBP will be obtained with a vital signs monitor
Change in average daytime ambulatory HR, and in average night-time ambulatory HR from baseline to the end of treatment. | from baseline to 3 months
  Daytime and nigh-time ambulatory HR will be obtained with 24hr ABPM
Change in BP variability defined as the coefficient of variation (SD/mean) of 24-hour ambulatory SBP, and of within-visit office SBP from baseline to the end of treatment. | from baseline to 3 months
  24hr ambulatory SBP will be obtained with 24hr ABPM
Change in Heart Rate (HR) variability defined as the coefficient of variation (SD/mean) of 24-hour ambulatory HR, and of within-visit office HR from baseline to the end of treatment. | from baseline to 3 months
  24hr ambulatory HR will be obtained with 24hr ABPM
Occurrence of a serious adverse event (SAE), fatal or non-fatal, within 3 months. | from baseline to 3 months
  SAEs will be collected through patient interviews, reporting and monitoring
The occurrence of a major cardiovascular event (MACE), including myocardial infarction (MI), stroke, and cardiovascular-related mortality within 3 months. | from baseline to 3 months
  MACE will be collected through patient interviews, reporting and monitoring
Change in Quality of life between baseline and the end of the treatment (3 months) using the EuroQol Visual Analogue score (0-100), and the EuroQol 5 Dimension (EQ5D) quality of life (QoL) questions. | from baseline to 3 months
  EQ-5D-5L questionnaire
Change in sleep quality between baseline and the end of the treatment using the Insomnia Severity Index (ISI), a 7-item questionnaire with each question allowing responses on a 5-point Likert scale from 0-4. Responses summed to give an overall score of 0 | from baseline to 3 months
  ISI questionnaires
Adherence to trial therapy, assessed as the proportion of days out of total days in follow-up when therapy was self-administered, and the average daily duration of self-administered therapy over the 3 months of follow-up (90 days). | from baseline to 3 months
  Study log-book

CONTACTS AND LOCATIONS:
Overall Officials: Ajay K Gupta, Principal Investigator — Queen Mary University of London
Locations (1):
- Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
On publication of findings relevant anonymized dataset will be made available to benefit researchers with justifiable reasons

REFERENCES:
- [Background] Markle W, M. Fisher, and R. Smego. Understanding Global Health. Economics and Global Health. 2007.
- [Background] Williams B, Mancia G, Spiering W, Agabiti Rosei E, Azizi M, Burnier M, Clement DL, Coca A, de Simone G, Dominiczak A, Kahan T, Mahfoud F, Redon J, Ruilope L, Zanchetti A, Kerins M, Kjeldsen SE, Kreutz R, Laurent S, Lip GYH, McManus R, Narkiewicz K, Ruschitzka F, Schmieder RE, Shlyakhto E, Tsioufis C, Aboyans V, Desormais I; ESC Scientific Document Group. 2018 ESC/ESH Guidelines for the management of arterial hypertension. Eur Heart J. 2018 Sep 1;39(33):3021-3104. doi: 10.1093/eurheartj/ehy339. No abstract available. PMID 30165516
- [Background] England PH. Health matters: preventing cardiovascular disease 2019.
- [Background] Foundation BH. BHF Coronavirus and Heart & Circulatory Disease Statistics. 2020.
- [Background] Egan BM, Kjeldsen SE, Grassi G, Esler M, Mancia G. The global burden of hypertension exceeds 1.4 billion people: should a systolic blood pressure target below 130 become the universal standard? J Hypertens. 2019 Jun;37(6):1148-1153. doi: 10.1097/HJH.0000000000002021. PMID 30624370
- [Background] England PH. Hypertension prevalence estimates in England. 2017;2020.
- [Background] England PH. Tackling high blood pressure From evidence into action. 2014.
- [Background] Achelrod D, Wenzel U, Frey S. Systematic review and meta-analysis of the prevalence of resistant hypertension in treated hypertensive populations. Am J Hypertens. 2015 Mar;28(3):355-61. doi: 10.1093/ajh/hpu151. Epub 2014 Aug 25. PMID 25156625
- [Background] Abegaz TM, Shehab A, Gebreyohannes EA, Bhagavathula AS, Elnour AA. Nonadherence to antihypertensive drugs: A systematic review and meta-analysis. Medicine (Baltimore). 2017 Jan;96(4):e5641. doi: 10.1097/MD.0000000000005641. PMID 28121920
- [Background] Carey RM, Calhoun DA, Bakris GL, Brook RD, Daugherty SL, Dennison-Himmelfarb CR, Egan BM, Flack JM, Gidding SS, Judd E, Lackland DT, Laffer CL, Newton-Cheh C, Smith SM, Taler SJ, Textor SC, Turan TN, White WB; American Heart Association Professional/Public Education and Publications Committee of the Council on Hypertension; Council on Cardiovascular and Stroke Nursing; Council on Clinical Cardiology; Council on Genomic and Precision Medicine; Council on Peripheral Vascular Disease; Council on Quality of Care and Outcomes Research; and Stroke Council. Resistant Hypertension: Detection, Evaluation, and Management: A Scientific Statement From the American Heart Association. Hypertension. 2018 Nov;72(5):e53-e90. doi: 10.1161/HYP.0000000000000084. PMID 30354828
- [Background] Dahal K, Khan M, Siddiqui N, Mina G, Katikaneni P, Modi K, Azrin M, Lee J. Renal Denervation in the Management of Hypertension: A Meta-Analysis of Sham-Controlled Trials. Cardiovasc Revasc Med. 2020 Apr;21(4):532-537. doi: 10.1016/j.carrev.2019.07.012. Epub 2019 Jul 26. PMID 31420197
- [Background] Gupta A, Prince M, Bob-Manuel T, Jenkins JS. Renal denervation: Alternative treatment options for hypertension? Prog Cardiovasc Dis. 2020 Jan-Feb;63(1):51-57. doi: 10.1016/j.pcad.2019.12.007. Epub 2019 Dec 27. PMID 31884099
- [Background] Azizi M, Schmieder RE, Mahfoud F, Weber MA, Daemen J, Lobo MD, Sharp ASP, Bloch MJ, Basile J, Wang Y, Saxena M, Lurz P, Rader F, Sayer J, Fisher NDL, Fouassier D, Barman NC, Reeve-Stoffer H, McClure C, Kirtane AJ; RADIANCE-HTN Investigators. Six-Month Results of Treatment-Blinded Medication Titration for Hypertension Control After Randomization to Endovascular Ultrasound Renal Denervation or a Sham Procedure in the RADIANCE-HTN SOLO Trial. Circulation. 2019 May 28;139(22):2542-2553. doi: 10.1161/CIRCULATIONAHA.119.040451. Epub 2019 Mar 17. PMID 30880441
- [Background] Kandzari DE, Bohm M, Mahfoud F, Townsend RR, Weber MA, Pocock S, Tsioufis K, Tousoulis D, Choi JW, East C, Brar S, Cohen SA, Fahy M, Pilcher G, Kario K; SPYRAL HTN-ON MED Trial Investigators. Effect of renal denervation on blood pressure in the presence of antihypertensive drugs: 6-month efficacy and safety results from the SPYRAL HTN-ON MED proof-of-concept randomised trial. Lancet. 2018 Jun 9;391(10137):2346-2355. doi: 10.1016/S0140-6736(18)30951-6. Epub 2018 May 23. PMID 29803589
- [Background] Clancy JA, Mary DA, Witte KK, Greenwood JP, Deuchars SA, Deuchars J. Non-invasive vagus nerve stimulation in healthy humans reduces sympathetic nerve activity. Brain Stimul. 2014 Nov-Dec;7(6):871-7. doi: 10.1016/j.brs.2014.07.031. Epub 2014 Jul 16. PMID 25164906
- [Background] Bretherton B, Atkinson L, Murray A, Clancy J, Deuchars S, Deuchars J. Effects of transcutaneous vagus nerve stimulation in individuals aged 55 years or above: potential benefits of daily stimulation. Aging (Albany NY). 2019 Jul 30;11(14):4836-4857. doi: 10.18632/aging.102074. PMID 31358702
- [Background] Redgrave J, Day D, Leung H, Laud PJ, Ali A, Lindert R, Majid A. Safety and tolerability of Transcutaneous Vagus Nerve stimulation in humans; a systematic review. Brain Stimul. 2018 Nov-Dec;11(6):1225-1238. doi: 10.1016/j.brs.2018.08.010. Epub 2018 Aug 23. PMID 30217648
- [Background] Ettehad D, Emdin CA, Kiran A, Anderson SG, Callender T, Emberson J, Chalmers J, Rodgers A, Rahimi K. Blood pressure lowering for prevention of cardiovascular disease and death: a systematic review and meta-analysis. Lancet. 2016 Mar 5;387(10022):957-967. doi: 10.1016/S0140-6736(15)01225-8. Epub 2015 Dec 24. PMID 26724178
- [Background] van Bilsen M, Patel HC, Bauersachs J, Bohm M, Borggrefe M, Brutsaert D, Coats AJS, de Boer RA, de Keulenaer GW, Filippatos GS, Floras J, Grassi G, Jankowska EA, Kornet L, Lunde IG, Maack C, Mahfoud F, Pollesello P, Ponikowski P, Ruschitzka F, Sabbah HN, Schultz HD, Seferovic P, Slart RHJA, Taggart P, Tocchetti CG, Van Laake LW, Zannad F, Heymans S, Lyon AR. The autonomic nervous system as a therapeutic target in heart failure: a scientific position statement from the Translational Research Committee of the Heart Failure Association of the European Society of Cardiology. Eur J Heart Fail. 2017 Nov;19(11):1361-1378. doi: 10.1002/ejhf.921. Epub 2017 Sep 26. PMID 28949064
- [Background] Rahimi K. Blood pressure reduction - lower really is better. European Society of Cardiology. 2020.
- [Background] Mueller ST, Piper BJ. The Psychology Experiment Building Language (PEBL) and PEBL Test Battery. J Neurosci Methods. 2014 Jan 30;222:250-9. doi: 10.1016/j.jneumeth.2013.10.024. Epub 2013 Nov 20. PMID 24269254
- [Background] Voils CI, Maciejewski ML, Hoyle RH, Reeve BB, Gallagher P, Bryson CL, Yancy WS Jr. Initial validation of a self-report measure of the extent of and reasons for medication nonadherence. Med Care. 2012 Dec;50(12):1013-9. doi: 10.1097/MLR.0b013e318269e121. PMID 22922431
- [Background] Bang H, Ni L, Davis CE. Assessment of blinding in clinical trials. Control Clin Trials. 2004 Apr;25(2):143-56. doi: 10.1016/j.cct.2003.10.016. PMID 15020033
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246